CLINICAL TRIAL: NCT05539443
Title: Telehealth-Enhanced Assessment and Management After Stroke-Blood Pressure
Acronym: TEAMS-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00085596; PLACER-02020C3-21070 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2022-08-11; First posted 2022-09-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-07

CONDITIONS: Hypertension Secondary
Keywords: Hypertension; Hypertension after stroke
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Clinic Management (ICM) (Experimental)
  Interventions: Behavioral: Intensive Clinic Management (ICM)
- Intensive tailored telehealth management (ITTM) (Experimental)
  Interventions: Behavioral: Intensive tailored telehealth management (ITTM)

INTERVENTIONS:
Behavioral: Intensive Clinic Management (ICM) — An in-person clinic management based on the intervention tested among stroke patients in the Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis (SAMMPRIS) trial
  Arms: Intensive Clinic Management (ICM)
Behavioral: Intensive tailored telehealth management (ITTM) — A remote-monitoring blood pressure (BP) management strategy incorporating individualized lifestyle coaching and care planning based on the HyperLink telehealth management trial
  Arms: Intensive tailored telehealth management (ITTM)

SUMMARY:
TEAMS-BP is a multicenter, participant-randomized controlled trial designed to compare the effectiveness of Intensive Tailored Telehealth Monitoring (ITTM) versus Intensive Clinic Management (ICM) on Blood Pressure (BP) control and patient activation for BP management following stroke

DETAILED DESCRIPTION:
The Feasibility phase will allow for a period in which to pilot implementation and evaluation of all systems for data acquisition, clinical management, and collection of 3-month outcomes. The study uses a parallel, 2-arm design with 1-to-1 randomization to treatment group. Randomization will be performed at the participant level, stratified by center, age (18-74, 75+), and race (Black/African American, non-Black/African American).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke defined as acute brain, spinal cord, or retinal infarction based on objective evidence on imaging (such as a focal area of restricted diffusion on Magnetic Resonance Imaging [MRI]) in a defined vascular distribution or clinical evidence of focal ischemic injury based on symptoms persisting > 24 hours; or spontaneous hemorrhagic stroke defined as a focal collection of blood within the brain parenchyma that is non-traumatic and identified by brain computed tomography (CT) or brain MRI
* Age ≥18 years
* Discharged directly home from acute care or inpatient rehabilitation
* SBP>130 at the post-acute clinic visit (within 21 days of discharge) & at Study Visit 1 (within 31 days of discharge)
* Able to read and understand English or Spanish
* Have access to a functioning smartphone or tablet with broadband access (required for the intervention)
* Willing to install and use a study-compatible physical activity monitoring application on their smartphone or smartphone of a qualifying caregiver
* Stated agreement to participate in either intervention to which they are assigned and attend all required study visits
* Consent to receiving Short Message Service (SMS) required as part of the study interventions
* Provision of a signed and dated informed consent form

Exclusion Criteria:

* Subdural hematoma or subarachnoid hemorrhage
* Current participation in another stroke clinical trial precluding dual enrollment
* Presence of terminal illness, such as cancer, that limits life expectancy to <1 year
* Diagnosis of end-stage renal disease defined as permanent kidney dysfunction requiring the use of hemodialysis or peritoneal dialysis
* Pregnancy, lactation or planning to become pregnant
* Late-stage Alzheimer's disease or related dementia
* Transitioned to a facility such as skilled nursing or long-term care prior to enrollment
* Any condition that in the opinion of the study investigator would preclude the participant from being able to safely participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with 3-month SBP control | 3 months

SECONDARY OUTCOMES:
Mean change in systolic blood pressure (SBP) at 3 months | Baseline, 3 month
  Defined as the SBP at baseline (Visit 1) subtracted from the SBP at 3 months (Visit 2).
Mean change in Partners in Health Scale (PIH) score at 3 months | Baseline, 3 month
  Each of the 11 items on the PIH have eight response options ranging from (0) very good to (8) very poor. To calculate the total PIH score, the raw score is summed and transformed to a range [0,100], with lower PIH scores indicating higher patient activation.
Proportion of participants eligible among those screened | 3 Month
Proportion of participants providing written informed consent among those eligible | Baseline
Proportion of participants attending both visits among those who are randomized in the study | 3 months
Systolic Blood Pressure Mean Value | 3 months
Proportion of respondents with top score in overall experience on the Research Participant Perception Survey (RPPS) | 3 months
  The overall experience (Overall Rating) is rated on a 10-point scale from 0 (Worst) to 10 (Best). The top score is for overall score includes all participants that responded 9 or 10.
Proportion of participants billed | 3 months
  Proportion of participants for which coaching or remote physiologic monitoring services were billed (at any point during the study) using Current Procedural Terminology (CPT) billing codes.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Bushnell, MD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT05539443/ICF_000.pdf